CLINICAL TRIAL: NCT00290693
Title: A Multicenter Phase II Study of Capecitabine and Docetaxel for Previously Treated Pancreatic Cancer Patients "CapTere"
Brief Title: Capecitabine and Docetaxel in Treating Patients With Recurrent or Progressive Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20030652; SCCC-2003099 (Other: UM/Sylvester Comprehensive Cancer Center); WIRB-20051007 (Other: Western Institutional Review Board); AVENTIS-14056 (Other: Aventis)
Record Dates: First submitted 2006-02-09; First posted 2006-02-13 (Estimated); Results first posted 2013-05-13 (Estimated); Last update posted 2017-12-02 (Actual); Status verified 2017-10

CONDITIONS: Pancreatic Cancer
Keywords: recurrent pancreatic cancer; adenocarcinoma of the pancreas; stage IV pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Capecitabine; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CapTere (Capecitabine + Docetaxel) (Experimental): Capecitabine + Docetaxel (Taxotere)
  Interventions: Drug: Capecitabine; Drug: Docetaxel

INTERVENTIONS:
Drug: Capecitabine — Orally, 1600mg/m2/day given as (800mg/m2 BID), Days 1 through 14 of 21-day cycle
  Other Names: Xeloda
Drug: Docetaxel — 30 mg/m2, IV, days 1 and 8 every 3 weeks
  Other Names: Taxotere

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as capecitabine and docetaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving capecitabine together with docetaxel works in treating patients with recurrent or progressive metastatic pancreatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the overall (complete and partial) response rate in patients with recurrent or progressive metastatic pancreatic cancer treated with capecitabine and docetaxel.

Secondary

* Determine the overall and progression-free survival of patients treated with the chemotherapy combination.
* Determine the duration of response (complete or partial) among patients who attain a response.
* Determine the frequency of patients having > 50% fall of CA19-9 from an initial level of > 100 U/mL in association with treatment with this regimen.
* Evaluate the toxicity associated with the administration of the combination in these patients.

OUTLINE: This is a multicenter, open-label, nonrandomized study.

Patients receive oral capecitabine twice daily on days 1-14 and docetaxel IV over 1 hour on days 1 and 8. Treatment repeats every 3 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months for up to 1 year.

PROJECTED ACCRUAL: A total of 45 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

1. Participants or their authorized legally acceptable representative must consent to be in the study and must have signed and dated an approved consent form which conforms to federal and institutional guidelines.
2. Patients must be 18 years or older.
3. Participants must have recurrence or progression of histologically or cytologically documented pancreatic adenocarcinoma. Re-documentation of tumor histology or cytology prior to protocol therapy is not required if documented tumor was confirmed prior to initial therapy.
4. Patients must have metastatic disease.
5. Patients with metastatic disease to the brain if they have received radiation therapy or are stable, and are not receiving steroids or anticonvulsants.
6. Participants must have received one prior gemcitabine based chemotherapy regimen (with or without radiation therapy). Participants must be 3 weeks or more beyond completion of prior chemotherapy (30 days beyond any experimental agent) and show recovery from toxicity to within the eligibility parameters of this protocol.
7. Radiation for palliation and of the primary tumor must have been completed at least four weeks prior to initiation of protocol therapy.
8. Patients must have measurable tumor by Response Evaluation Criteria in Solid Tumors (RECIST) (Therasse et al, 2000). Measurable disease includes any lesion ≥ 1 cm by spiral CT or ≥ 2 cm by non-spiral CT in longest diameter which can be repetitively assessed by radiographic measurement or any lesion ≥ 2 cm in longest diameter which can be repetitively assessed by physical examination. Positive bone scans, osteoblastic or osteolytic bone lesions, pleural effusions and positive bone marrow biopsies are not considered acceptable as either measurable or evaluable lesions.
9. Participants must have Eastern Cooperative Oncology Group (ECOG) Performance Status Score of 0,1, or 2.
10. Females of reproductive potential must not plan on conceiving children during the treatment period and must agree to use an effective medically accepted form of contraception. Patients will agree to continue contraception for 60 days from the date of the last study drug administration.
11. Required initial laboratory data:

    * Granulocytes ≥ 1,500/µl
    * Platelets ≥ 100,000/µl
    * Hg ≥ 8.0 g/dL
    * Creatinine ≤ 2.0 mg/dL
    * Creatine Clearance >30 ml/min as calculated with Cockroft-Gault equation
    * Bilirubin ≤ Upper Limits of Normal (ULN)
    * Pregnancy test for females with child-bearing potential: Negative within 7 days of starting protocol
12. Transaminases (SGOT and/or SGPT) may be up to 2.5 x institutional upper limit of normal (ULN) if alkaline phosphatase is ≤ ULN, or alkaline phosphatase may be up to 4 x ULN if transaminases are ≤ ULN.

Exclusion Criteria:

1. Patient currently enrolled in another clinical trial.
2. Pregnant or breast feeding women. With the exception of post-menopausal or infertile women, a negative blood test for pregnancy is mandatory before entry on study. Fertile persons refusing to use contraceptives may not participate.
3. Participants may not have had capecitabine or docetaxel as part of prior therapy.
4. No concurrent clinically evident malignancy is allowed except inactive non-melanoma skin cancer, low grade low stage bladder carcinoma followed off therapy, treated in-situ cervical cancer or lobular neoplasia of the breast.
5. Participants with serious uncontrolled medical or psychiatric illness that would render chemotherapy unsafe are ineligible.
6. Pregnant or breast-feeding at the time of proposed study entry.
7. Clinical AIDS or known positive HIV serology.
8. Peripheral neuropathy > grade 1
9. Patients with a history of severe hypersensitivity reaction to drugs formulated with polysorbate 80 must be excluded.
10. Prior unanticipated severe reaction to fluoropyrimidine therapy, or known sensitivity to 5-fluorouracil.
11. Clinically significant cardiac disease (e.g. congestive heart failure, symptomatic coronary artery disease and cardiac arrhythmias not well controlled with medication) or myocardial infarction within the last 12 months.
12. Lack of physical integrity of the upper gastrointestinal tract or malabsorption syndrome.
13. Major Surgery within 4 weeks of the start of study treatment, without complete recovery.
14. Unwillingness to participate or inability to comply with the protocol for the duration of the study.
15. Patients with impaired renal function (estimated creatinine clearance < 30 ml/min as calculated by the Cockroft-Gault Equation).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2004-07 (Actual); Primary Completion 2008-08 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Caio Max S. Rocha Lima, MD, Principal Investigator — University of Miami
Locations (3):
- United States (3):
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - Mount Sinai Comprehensive Cancer Center at Mount Sinai Medical Center, Miami Beach, Florida

REFERENCES:
- [Result] Soares HP, Bayraktar S, Blaya M, Lopes G, Merchan J, Macintyre J, Mayo C, Green MR, Silva O, Levi J, Walker G, Rocha-Lima CM. A phase II study of capecitabine plus docetaxel in gemcitabine-pretreated metastatic pancreatic cancer patients: CapTere. Cancer Chemother Pharmacol. 2014 Apr;73(4):839-45. doi: 10.1007/s00280-014-2414-z. Epub 2014 Feb 23. PMID 24562589

RESULTS

PARTICIPANT FLOW:
Groups:
- CapTere (Capecitabine + Docetaxel): Docetaxel : 30 mg/m2, IV, days 1 and 8 every 3 weeks
  Capecitabine : Orally, 1600mg/m2/day given as (800mg/m2 BID), Days 1 through 14 of 21-day cycle
Period: Overall Study
Arm/Group | CapTere (Capecitabine + Docetaxel)
Started | 45
Completed | 43
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: The 43 study participants who completed baseline assessments and received at least one dose of protocol therapy.
Groups:
- CapTere (Capecitabine + Docetaxel): * Docetaxel : 30 mg/m2, IV, days 1 and 8 every 3 weeks
  * Capecitabine : Orally, 1600mg/m2/day given as (800mg/m2 BID), Days 1 through 14 of 21-day cycle
Arm/Group | CapTere (Capecitabine + Docetaxel)
Number analyzed (Participants) | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 21
  >=65 years | 22
Age, Continuous [Median (Full Range); unit: years] | 64.4 [44 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 22
Region of Enrollment [Number; unit: participants]
  United States | 43

OUTCOME MEASURES:

1. Primary Outcome: Rate of Participants Achieving Complete Response or Partial Response to Therapy.
Description: Rate of participants achieving complete response (CR) or partial response (PR) to Captere therapy according to RECIST criteria v 1.0. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions.
Time Frame: Up to 1 year
Population: Number of participants evaluable for response, that is, who completed at least one cycle of protocol therapy.
Measure: Number; unit: participants
Arm/Group | CapTere (Capecitabine + Docetaxel)
Number analyzed (Participants) | 42
participants
  Partial Response (PR) >= 2 cycles | 6
  Stable Disease (SD), >= 2 cycles | 25
  Complete Response (CR), >= 2 cycles | 0

2. Secondary Outcome: Overall Surival (OS)
Description: Overall survival is measured from the time from date of initial protocol therapy to date of death. In the absence of confirmation of death, survival time will be censored to last date of follow-up.
Time Frame: Up to 1 year
Population: Number of participants who completed at least one cycle of protocol therapy.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | CapTere (Capecitabine + Docetaxel)
Number analyzed (Participants) | 42
months | 5.3 [4.3 to 8.6]

3. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival (PFS) is measured the time from the start of protocol therapy to disease progression or death from any cause. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Up to 1 year
Population: Number of participants who completed at least one cycle of protocol therapy.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | CapTere (Capecitabine + Docetaxel)
Number analyzed (Participants) | 42
months | 3.7 [2.1 to 4.3]

4. Secondary Outcome: Rate of Participants Achieving a 50% or More Reduction in CA 19-9 Levels
Description: Rate of participants achieving a 50% or more reduction in CA 19-9 levels after receiving protocol therapy. Baseline CA-19-9 will be compared to the lowest recorded value on patients receiving therapy on protocol. A 50% drop in CA 19-9 in patients with baseline levels above 100 U/ml will be recorded as a CA 19-9 response if the > 50% drop can be confirmed with at least one more CA 19-9 level thereafter with > 50% drop compared to baseline.
Time Frame: Up to 1 year
Population: Participants who had available baseline CA19-9 levels above 100 U/ml.
Measure: Number; unit: percentage of participants
Arm/Group | CapTere (Capecitabine + Docetaxel)
Number analyzed (Participants) | 31
percentage of participants | 35.48

5. Secondary Outcome: Number of Study Participants Experiencing Toxicity After Receiving Protocol Therapy
Description: Number of study participants experiencing toxicity (serious adverse events or adverse events). Study participants assessed for this outcome measure must have received at least one dose of protocol therapy. Toxicity assessed according to Common Terminology Criteria for Adverse Events v3.0 (CTCAE).
Time Frame: Up to 1 year
Population: Study participants who received at least one dose of protocol therapy.
Measure: Number; unit: participants
Arm/Group | CapTere (Capecitabine + Docetaxel)
Number analyzed (Participants) | 43
participants | 38

ADVERSE EVENTS:
Description: Adverse events reported for the 43 participants receiving at least one dose of protocol therapy.
Arm/Group | CapTere (Capecitabine + Docetaxel)
All-Cause Mortality (participants affected / at risk) | 42/43
Serious Adverse Events (participants affected / at risk) | 25/43
Other Adverse Events (participants affected / at risk) | 20/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CapTere (Capecitabine + Docetaxel) (N=43)
Fatigue (General disorders) | 5 (5)
Hand and Foot Syndrome (Vascular disorders) | 6 (6)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Mucositis (Infections and infestations) | 2 (2)
Neuropathy (Nervous system disorders) | 1 (2)
Infection (Infections and infestations) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1)
Pleural Effusions (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nausea (Skin and subcutaneous tissue disorders) | 3 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CapTere (Capecitabine + Docetaxel) (N=43)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Neuropathy (Nervous system disorders) | 2 (2)
Mucositis (Infections and infestations) | 2 (2)
Hepatotoxicity (Hepatobiliary disorders) | 1 (1)
Hand and foot syndrome (Vascular disorders) | 5 (5)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes